CLINICAL TRIAL: NCT01560325
Title: Phase I Clinical Trial to Assess the Safety and Pharmacokinetic Profile of CKD-516 Inj. Administered on A Twice-Weekly Schedule in Patients With Advanced Solid Cancers Failed to Standard Therapy
Brief Title: Safety Study of Increasing Doses of CKD-516 in Patients With Advanced Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 127ASC12A
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Solid Tumor, Tubulin inhibitor
MeSH Terms: interventions — N-(4-(3-(1H-1,2,4-triazol-1-yl)-4-(3,4,5-trimethoxybenzoyl)phenyl)thiazol-2-yl)-2-amino-3-methylbutanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CKD-516 inj. (Experimental): CKD-516 Inj, 3.3~13mg/m2/day, D1, 4, 8, 11 every 3 weeks
  Interventions: Drug: CKD-516 inj.

INTERVENTIONS:
Drug: CKD-516 inj. — CKD-516: 3.3~13mg/m2/day
  Other Names: CKD-516

SUMMARY:
A phase I study is conducted to determine the maximum tolerated dose (MTD), dose limiting toxicity (DLT), safety and pharmacokinetics (PK) profile of a single agent CKD-516 injection on twice-weekly schedule in patients with advanced solid cancers failed to standard therapy. The usefulness of the this regimen is evaluated by response rate, progression free survival and vascular disruption effect by Dynamic Contrast-Enhanced MRI (DCE-MRI) or DWI.

DETAILED DESCRIPTION:
This is an open label, dose escalation study. Patients receive CKD-516 IV over 30 minutes on day 1, 4, 8, 11 every 3 weeks in the absence of unacceptable toxicity or disease progression. Cohorts of 3~6 patients receive escalating doses of CKD-516 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 20~75 years
* Histologically or cytologically confirmed solid tumors that have failed to standard therapy or for which no life prolonging treatment exists
* ECOG PS 0-2
* Life expectancy 12 weeks
* Hematopoietic: ANC ≥ 1,500/mm3, Platelet ≥ 100,000/mm3, Hemoglobin ≥ 9.0g/dL, Prothrombin time, Activated partial thromboplastin time: normal range
* Hepatic: total bilirubin ≤ 1.5×ULN(except Gilbert's syndrome patients), AST, ALT ≤ 3.0×ULN(AST, ALT ≤ 5.0×ULN in case of liver metastases)
* serum creatinine ≤ 1.5×ULN or Creatinine clearance ≥ 60 mL/min
* PT, APTT: normal range
* Signed a written informed consent

Exclusion Criteria:

* Brain or Leptomeningeal metastases
* History of Ischemic heart disease(e.g., myocardial infarction, unstable angina pectoris) or Clinically significant heart disease such as NYHA Class III and IV Congestive atrial arrhythmias, within 6 months prior to first dose of study drug
* Stable angina pectoris shown symptoms within 6 months prior to first dose of study durg, or Clinically significant abnormality on EKG or echocardiogram(e.g., LVEF < 50% or clinically significant heart wall abnormality or heart muscle damage)
* Cerebrovascular disease such as stroke
* Grade 2 or greater motor or sensory peripheral neuropathy
* Uncontrolled hypertension(greater than 150 mmHg systolic or 100 mmHg diastolic regardless of medication)
* acute infection or blooding tendencies that would preclude study compliance
* Serious vascular disease such as Aortic aneurysm
* Other psychiatric disorders or other conditions that would preclude study compliance
* Receiving anticoagulation with warfarin, heparin, etc.
* Receiving antitumor therapy(surgery, immunotherapy or chemotherapy) within 3 weeks prior to first dose of study drug(6 weeks for nitrosoureas and mitomycin C, 2 weeks for radiation therapy)
* Other concurrent antitumor therapy
* Patients with serious hypersensitivity history or allergy to CKD-516
* Pregnant or nursing, active serum pregnancy test. Fertile patients must use effective contraception
* Participation in a clinical trial within 4 weeks of first dose of study drug
* Patients judged to be inappropriate for this study by the investigator with other reasons

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
MTD, Maximum Tolerated Dose | up to 21days

SECONDARY OUTCOMES:
PK parameter of CKD-516 | 0(Pre-dose), 24hrs post dose (Day 1), 0, 0.5, 4, 8, 24hours post-dose(Day 11)
DLT, Dose-limiting Toxicity | up to 21days
ORR%, Objective response rate | up to 42weeks
Vascular disruption effect | 4hr, 24hr post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea